CLINICAL TRIAL: NCT03253432
Title: INTegrating Active Case-finding With Next-generation Sequencing for Diagnosis Through Electronic Medical Records (IN-TANDEM): Familial Hypercholesterolemia Pilot Study
Brief Title: IN-TANDEM Familial Hypercholesterolemia Pilot Study
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: The Familial Hypercholesterolemia Foundation (Other); Lancaster General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 826438
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Strata 0-0.05: Lowest probability of having familial hypercholesterolemia
  Interventions: Other: Genetic testing
- Strata 0.06-0.15: Second lowest probability of having familial hypercholesterolemia
  Interventions: Other: Genetic testing
- Strata 0.16-0.19: Moderate probability of having familial hypercholesterolemia
  Interventions: Other: Genetic testing
- Strata 0.20-0.34: Second highest probability of having familial hypercholesterolemia
  Interventions: Other: Genetic testing
- Strata greater than or equal to 35: Highest probability of having familial hypercholesterolemia
  Interventions: Other: Genetic testing

INTERVENTIONS:
Other: Genetic testing — Targeted next-generation sequencing for familial hypercholesterolemia causative mutations

SUMMARY:
The purpose of this study is to validate the use of the FH Foundation FIND FH® Algorithm as a clinical decision support tool. FIND FH (Flag/Identify/Network/Engage) is a national initiative that utilizes machine learning and data mining techniques to identify individuals whose profiles are consistent with FH patients. The algorithm will be tested in adults with at least one cardiovascular comorbidity. Study subjects will be asked to provide either a saliva, buccal or venous blood sample for DNA and biomarker analysis

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* At least one cardiovascular co-morbidity or receiving treatment for a cardiovascular comorbidity
* Algorithm score 0-1
* Most recent encounter with a provider within five years of query date

Exclusion Criteria:

* Any medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study, or confound study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Randomly selected patients from University of Pennsylvania and Lancaster General Hospital with at least 1 cardiovascular comorbidity seen at hospital within the past five years.
Sampling Method: Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

PRIMARY OUTCOMES:
Likelihood of having FH-causing mutation | 12 months
  Proportion of subjects with causative mutation in higher algorithm score groups

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with other investigators
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: De-identified data will be shared at end of study after database lock
Access Criteria: Research team

REFERENCES:
- [Derived] Qureshi N, Da Silva MLR, Abdul-Hamid H, Weng SF, Kai J, Leonardi-Bee J. Strategies for screening for familial hypercholesterolaemia in primary care and other community settings. Cochrane Database Syst Rev. 2021 Oct 7;10(10):CD012985. doi: 10.1002/14651858.CD012985.pub2. PMID 34617591